CLINICAL TRIAL: NCT03227822
Title: Short Spot Versus Long Lesion Stenting as Best Treatment for Extensive Occlusive SFA Disease; a Pilot Study
Brief Title: Short Spot Versus Long Lesion Stenting as Best Treatment for Extensive Occlusive SFA Disease
Acronym: STRONG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to include the number of patients
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Marc van Sambeek, MD, PhD, vascular surgeon, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STRONG SFA study; NL43610.060.13 (Registry Identifier: NL43610.060.13)
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short spot stenting (Experimental): Short spot stenting
  Interventions: Procedure: Short spot stenting
- Long lesion stenting (Experimental): Long lesion stenting
  Interventions: Procedure: Long lesion stenting

INTERVENTIONS:
Procedure: Short spot stenting
  Arms: Short spot stenting
Procedure: Long lesion stenting
  Arms: Long lesion stenting

SUMMARY:
Since the length of lesion seems to be negatively associated with stent patency due to restenosis, it is thought that the efficacy of treatment in patients with multiple (> 1) short (focal; > 1 and < 5 cm) SFA lesions can be improved by spot stenting as compared to the use of one long stent. This study proposes to evaluate the endovascular treatment for patients with SFA lesions by comparing two strategies for patients with extensive occlusive SFA disease; 1) short spot (SS) stenting or 2) long lesion (LL) stenting.

ELIGIBILITY:
Inclusion Criteria:

* PAOD (ABI <0.90 and/or a decline of >0.15 after exercise test), Rutherford category 2, 3 or 4
* Multiple (>1) short (focal; >1 and < 5 cm) significant stenoses (≥ 50%) and/or occlusions in the superficial femoral artery
* Eligible for endovascular treatment via short spot stenting and via long lesion stenting according to international guidelines
* Unilateral occlusive disease
* Age ≥ 18

Exclusion Criteria:

* Patients with PAOD Rutherford category 5 and 6
* Impaired inflow due to significant lesions in the arteries proximal to the SFA intended to treat
* Bilateral lesions with treatment indication
* Contra-indication for anticoagulant therapy
* Renal insufficiency (MDRD < 50 ml/min)
* Life expectancy < 6 months
* Known contrast allergy
* Pregnancy
* Unable to complete a questionnaire in the home language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02-01 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
absence of binary restenosis (≥ 50% re-obstruction) of the target lesion without interval clinically driven reintervention | 1 year